CLINICAL TRIAL: NCT04431167
Title: Healthy Lifestyle Intervention in Patients with Systemic Lupus Erythematosus with High Cardiovascular Risk: the Living Well with Lupus Study
Brief Title: Healthy Lifestyle Intervention in Patients with Systemic Lupus Erythematosus: the Living Well with Lupus Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Living well with lupus Study
Record Dates: First submitted 2020-02-18; First posted 2020-06-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Life style; Behavioral intervention; Cardiovascular risk; Life quality
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Experimental group and no intervention group (usual care group)
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for performing the blood flow measurement will be blinded to the allocation of groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Living well with Lupus Group (Experimental): A newly developed intervention focused on promoting lifestyle change through recommendations for structured and unstructured physical activity and healthy eating.
  Interventions: Behavioral: Living well with Lupus
- Usual Care Group (No Intervention): This group will receive all regular medical care and advice healthy

INTERVENTIONS:
Behavioral: Living well with Lupus — The lifestyle change intervention will involve two constructs: increasing the level of physical activity and improving eating habits, each with its own specific domains and goals. It will be based on a structured program of physical exercises and selection of individualized goals in the domains of transportation, leisure and work to reduce sedentary behavior with the aim of increasing the level of physical activity, as well as establishing changes in dietary aspects, involving consumption domains, structure, behavior and eating attitude using nutritional counseling techniques.
  Arms: Living well with Lupus Group

SUMMARY:
This research program aims to investigate the clinical, physiological, metabolic and molecular effects of lifestyle change in patients with systemic lupus erythematosus with high cardiovascular risk. This 6-month parallel-group randomized controlled trial aims to investigate the feasibility and efficacy of a newly developed lifestyle change intervention - through recommendations for structured and unstructured physical activity and healthy eating - on increasing physical activity level and improving eating habits. Potential effects of the intervention on cardiovascular and cardiometabolic risk factors, health-related quality of life, symptoms of anxiety and depression, sleep quality and immune function will be investigated. Gold-standard techniques and a variety of analyses will be performed to access the potential mechanisms involved in response to this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 65 years old diagnosed with systemic lupus erythematosus
* one or more high cardiovascular risk factors
* SLEDAI score ≤ 4
* Treatment with prednisone at a dosage <10 mg/d and treatment with hydroxychloroquine in a stable dose

Exclusion Criteria:

* another rheumatic diseases (except for secondary Sjogren's syndrome)
* participation in structured exercise training programs and/or prescriptive diets
* illiterate or with diagnosed cognitive disorders or musculoskeletal impairments that potentially compromise understanding and participation in the intervention

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants will be eligible
Enrollment: 80 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Risk cardiovascular score | 6 months
  assessed by measures of five standard variables (HDL cholesterol, triglycerides, fasting blood glucose, waist circumference and blood pressure - average of systolic and diastolic blood pressures). Z-score = [(50 - HDL cholesterol)/sd + (triglycerides - 150)/ sd] + [(fasting blood glucose - 100)/ sd] + [(waist circumference - 88)/ sd] + [(blood pressure - 115)/ sd]. Higher score values represent higher risk. *sd: standard deviation. Higher Z-score represent higher risk.

SECONDARY OUTCOMES:
Body mass index (BMI) | 6 months
  assessed by weight (kg) and height (m) that will be combined to report BMI in kg/m^2
Waist circumference (cm) | 6 months
  assessed by measuring tape positioned at the midpoint between the last floating vertebra and the iliac crest.
Total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides | 6 months
  assessed by blood sample analysis and combined to determine lipid profile
Insulin sensitivity | 6 months
  assessed by oral glucose tolerance test (OGTT)
Systolic and Diastolic blood pressure | 6 months
  assessed by auscultatory method with mercury sphygmomanometer
Physical activity level | 6 months
  assessed by thigh-mounted accelerometer (ActivPAL™ micro)
Food consumption | 6 months
  assessed by three 24-hour food recall in non-consecutive days (being one of the days on the weekend)
Visceral fat | 6 months
  assessed by tomography
Peak oxygen consumption, as assessed by a cardiopulmonary exercise test | 6 months
Endothelial function | 6 months
  assessed by flow-mediated vasodilatation (FMD)
Disease activity | 6 months
  The activity of the disease, which will be impaired by safety, will be assessed by the presence of anti-dsDNA, using the ELISA technique and confirmation by indirect immunofluorescence in Crithidia luciliae and assessed by the questionnaire Systemic lupus erythematosus disease activity index 2000 (SLEDAI-2000). Total score ranges from 0 to 105. Higher scores represent higher disease activity.
Damage index | 6 months
  assessed by Systemic Lupus International Collaborating Clinics/ American College of Rheumatology - Damage Index. Total score range from 0 (no damage) to 46 (maximum damage).
Global health status | 6 months
  assessed by the Visual Analogic Scale (0 and 10 scale). Higher values represent worst global health status.
Patients' perceptions of the intervention | 6 months
  assessed by focus group. A semi-structured script composed of open questions about intervention positive and negative points, barriers for physical activity practice and changes in food consumption, perceptions of health improvement or worsening (physical and psychological aspects), well-being, motivation to maintain the changes made, perspectives regarding health and disease.
Quality of Life assesment assessed by the Short-Form Health Survey-36 (SF36) [followed by its scale information in the Description] | 6 months
  maximum score is 100, with higher scores representing better life quality
Quality of Life assessed by Systemic Lupus Erythematosus Quality of Life Questionnaire ( SLEQOL) [followed by its scale information in the Description] | 6 months
  score ranges from 40 to 280 with higher scores represent worst life quality.
Physical functioning assessed by Timed-Stands | 6 months
  evaluates the maximum number of stand-ups that a subject could perform from a standard height (i.e., 45 cm) armless chair within 30 s
Physical functioning assessed by Timed Up-and-Go | 6 months
  evaluates the time required for the subject to rise from a standard arm chair, walk towards a line drawn on the floor three meters away, turn, return, and sit back down again
Physical functioning assessed by handgrip test | 6 months
  Patients will be instructed to squeeze the dynamometer as hard as possible
Fatigue | 6 months
  assessed by Fatigue Scale (FACIT). The final score can vary from 0 to 52, where higher final score representing higher level of fatigue.
Anxiety | 6 months
  assessed by sub-scale of Hospital Anxiety and Depression Scale (HADS), called HADS-A. Total score ranges from 0 to 21. Where higher final score representing higher level.
Depression | 6 months
  assessed by sub-scale of Hospital Anxiety and Depression Scale (HADS), called HADS-D. Total score ranges from 0 to 21. Where higher final score representing higher level.
Sleep quality assessed by data obtained from Actigraph (Actigraph GT3x) | 6 months
  Data from actigraph will come as these measures: Total Sleep Time (hours/day), Sleep Efficiency (%), Sleep Onset Latency (min), and Wake After Sleep Onset (min), and this data will be considered to determine the sleep quality.
C-reactive protein (PCR) | 6 months
  assessed by analysis of blood sample
Erythrocyte sedimentation rate | 6 months
  assessed by analysis of blood sample
Inflammatory markers (blood biochemistry) | 6 months
  assessed by serum cytokines
Follow-up | Between 7 and 28 months after the completion of the intervention
  investigate the long-term effects of the intervention on maintenance of lifestyle behaviors and its effects on health

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
we can share the individual data of the participants if the request is reasonable

REFERENCES:
- [Derived] Caruso Mazzolani B, Infante Smaira F, Mendes Sieczkowska S, Romero M, C Santo Andre H, G Pasoto S, de Sa Pinto AL, Rodrigues Lima F, Braga Benatti F, Roschel H, Weber MB, Gualano B. Acceptability and impact of a lifestyle intervention for systemic lupus erythematosus: Qualitative analysis of living well with lupus study. Lupus. 2025 Apr;34(5):474-483. doi: 10.1177/09612033251326986. Epub 2025 Mar 13. PMID 40083122
- [Derived] Sieczkowska SM, Mazzolani BC, Smaira FI, Romero M, Pasoto SG, de Sa Pinto AL, Lima FR, De Oliveira VR, Ueda S, Benatti FB, Roschel H, Gualano B. Effects of a lifestyle intervention on cardiovascular risk factors in systemic lupus erythematosus patients: The study "Living well with lupus". Clin Rheumatol. 2024 Mar;43(3):1003-1013. doi: 10.1007/s10067-024-06870-2. Epub 2024 Jan 27. PMID 38280124
- [Derived] Sieczkowska SM, Smaira FI, Mazzolani BC, Romero M, Pasoto SG, de Sa Pinto AL, Lima FR, De Oliveira VR, Ueda S, Benatti FB, Roschel H, Gualano B. A randomized controlled trial of an intervention promoting physical activity and healthy eating recommendations in systemic lupus erythematosus: the protocol study "Living Well with Lupus". Rheumatol Int. 2023 Oct;43(10):1799-1810. doi: 10.1007/s00296-023-05370-x. Epub 2023 Jun 24. PMID 37354245